CLINICAL TRIAL: NCT02003781
Title: Individualized Prevention Strategy for High Risk Patients in Cardiovascular Disease: Prospective Cohort Study (Cardiovascular and Metabolic Disease Etiology Research Center - HIgh Risk Cohort) CMERC-HI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0581
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: High Risk Cardiovascular Disease Patients
Keywords: cardiovascular disease; metabolic disease; high risk; prospective cohort
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, whole blood, urine, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiovascular disease: high risk cardiovascular disease patients and their relatives

SUMMARY:
Set the prospective cohort (CMERC-HI) to study the known and novel etiologies and related factors for predicting clinical outcomes in Korean patients with high risk cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* high risk hypertension patients a. eGFR > 60 with one of target organ damages b. eGFR <= 60
* diabetes mellitus with microalbumin ration (AC ratio >= 30mg/g)
* anuric ESRD patients on dialysis
* the relatives of acute myocardial infarction patients under 55 years old (men)/ 65 years old (women)
* atherosclerotic cardiovascular disease (abdominal aorta diameter ≥3 cm or ankle-brachial index <0.9, or carotid plaque or carotid intima-media thickness ≥0.9 mm, or asymptomatic old cerebrovascular accident, or >30% stenosis in at least one major coronary artery)
* rheumatoid arthritis patients aged > 40 years on MTX and steroid therapy
* atrial fibrillation patients with CHADS-VASc Score ≥ 1
* kidney transplant recipient at > 3 months after transplantation

Exclusion Criteria:

* acute myocardial infarction, acute coronary syndrome patients, symptomatic coronary artery disease or history of these diseases
* symptomatic peripheral artery disease, heart failure and history of these diseases
* desired life time under 6 months due to non-cardiovascular disease (e.g. cancer, sepsis)
* women with pregnancy or on nursing
* history of contrast allergy and related side effects
* within the first three months after transplantation
* acute renal allograft rejection

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: high risk cardiovascular disease patients and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-10; Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Prognosis of high risk cardiovascular disease | 10 year after recruting
  all-cause mortality, cardiovascular mortality, non-cardiovascular mortality
  new onset of acute myocardial infarction, acute coronary syndrome, heart failure, stroke, peripheral artery disease, hospitalization for revascularization and these disease

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Seo J, Lee CJ, Oh J, Lee SH, Kang SM, Park S. Large discrepancy between unobserved automated office blood pressure and ambulatory blood pressure in a high cardiovascular risk cohort. J Hypertens. 2019 Jan;37(1):42-49. doi: 10.1097/HJH.0000000000001868. PMID 30507862
- [Derived] Park S, Lee CJ, Jhee JH, Yun HR, Kim H, Jung SY, Kee YK, Yoon CY, Park JT, Kim HC, Han SH, Kang SW, Park S, Yoo TH. Extracellular Fluid Excess Is Significantly Associated With Coronary Artery Calcification in Patients With Chronic Kidney Disease. J Am Heart Assoc. 2018 Jun 30;7(13):e008935. doi: 10.1161/JAHA.118.008935. PMID 29960990
- [Derived] Joo WT, Lee CJ, Oh J, Kim IC, Lee SH, Kang SM, Kim HC, Park S, Youm Y. The Association between Social Network Betweenness and Coronary Calcium: A Baseline Study of Patients with a High Risk of Cardiovascular Disease. J Atheroscler Thromb. 2018 Feb 1;25(2):131-141. doi: 10.5551/jat.40469. Epub 2017 Jul 21. PMID 28740058
- [Derived] Oh J, Lee CJ, Kim IC, Lee SH, Kang SM, Choi D, Park S, Kario K. Association of Morning Hypertension Subtype With Vascular Target Organ Damage and Central Hemodynamics. J Am Heart Assoc. 2017 Feb 14;6(2):e005424. doi: 10.1161/JAHA.116.005424. PMID 28196818